CLINICAL TRIAL: NCT06345222
Title: Examining the Effect of Prolotherapy on Quality of Life and Painkiller Use in Patients With Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hakan Demirci, Professor, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAT 23/05
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: The Aim of This Research is to Investigate the Effect of Prolotherapy on Quality of Life and Painkiller Use in Patients With Chronic Knee Pain
MeSH Terms: interventions — Prolotherapy

STUDY DESIGN:
Intervention Model Description: Case control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolotherapy (Experimental): Patients to whom prolotherapy treatment applied (n=32).
  Interventions: Procedure: Prolotherapy
- Control (Other): Patients to whom no prolotherapy applied. No intervention with their treatment (n=33).
  Interventions: Procedure: Prolotherapy

INTERVENTIONS:
Procedure: Prolotherapy — The "Modified Prolotherapy" technique was applied in the study and 0.5cc 5% Dextrose injection was applied per injection to the tendon entesis and/or tendon of the patient's non-rheumatic chronic, myoskeletal knee-induced, pain-inducing sensation. The follow-up period was determined as 1 month after the last injection. The ligaments to be injected within the scope of the research (context knee pain) were determined as Lateral Collateral Ligament (LCL), AnteroLateral Collateral Ligament (ALL), Medial Collateral Ligament (MCL), Pes Anserius and Patellar Ligament.

SUMMARY:
92 patients with a diagnosis of primary knee pain of unknown cause followed at the family medicine outpatient clinic and who met our exclusion criteria were invited to the study. When creating patient list, the examination of patients, interviews with patients, as well as their medical records and examinations were used. Patients were divided into two groups: prolotherapy (n=46) and control group (n=46) by simple randomization method. However, when the study started, 32 people in the prolotherapy group and 33 people in the control group of these patients participated in the study. Prior to the research, detailed information was provided about the research in the experimental and control groups and signed consent was obtained from all participants that they volunteered to participate in the research. 5% dectrose was applied to the prolotherapy group by injection method to the pain area. In the control group, existing medical treatments were continued and no injection procedure was performed. Before the research, all participants were evaluated with Case Report Form, Visual Analog Scale (VAS) and Quality of Life Scale Short Form (SF-36). The cases in the experimental and control groups were re-evaluated with the VAS and SF-36 scales at the first month.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffer from primary knee osteoarthritis

Exclusion Criteria:

* Inflammatory knee pain
* Cellulitis
* Septic arthritis
* Local abscess
* Bleeding disorders
* Patient on anticoagulant medication
* Patients allergic to dextrose
* Diabetes Mellitus
* breathing problems
* Electrolyte imbalance
* Kidney or liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
change in knee pain with prolotherapy application | 1 month
  Visual Analog Scale (VAS) scores determines pain relief. VAS scale use numbers from 0 to 10. A score of 0 means no pain, and 10 means the worst pain you have ever felt.
change in quality of life | 1 month
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.SF-36 Scale scores determines change in quality of life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Demirci, Professor, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on demand. Sharing data identifying patients is forbidden in Türkiye.